CLINICAL TRIAL: NCT01375972
Title: Randomized Phase II Trial of SP vs. GP in Advanced Biliary Cancer
Brief Title: Trial of S-1 Plus Cisplatin (SP) Versus Gemcitabine Plus Cisplatin (GP) in Advanced Biliary Tract Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_0803
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Metastatic Biliary Cancer
Keywords: biliary cancer; systemic chemotherapy; S-1; gemcitabine; cisplatin
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — S-1 plus cisplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP treatment (Experimental): S-1 plus cisplatin combination chemotherapy
  Interventions: Drug: S-1 plus cisplatin
- GP treatment (Active Comparator): Gemcitabine plus Cisplatin combination chemotherapy
  Interventions: Drug: Gemcitabine plus Cisplatin

INTERVENTIONS:
Drug: S-1 plus cisplatin — S-1 40 mg/m2 D1-D14 Cisplatin 60 mg/m2 D1 every 3 weeks
  Arms: SP treatment
Drug: Gemcitabine plus Cisplatin — Gemcitabine 1000 mg/m2 IV D1, D8 Cisplatin 60 mg/m2 IV D1 Every 3 weeks
  Arms: GP treatment

SUMMARY:
To select a better agent between S-1 or gemcitabine in combination with cisplatin for the conventional chemotherapy platform for future development in advanced Biliary Tract Adenocarcinoma (BTA), the investigators conduct a randomized phase II trial of S-1 and cisplatin (SP) versus gemcitabine and cisplatin (GP) as first line therapy in advanced BTA.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven biliary adenocarinoma
2. Age > 18
3. Evaluable disease
4. ECOG performance status of 2 or better
5. No prior exposure to chemotherapy, but adjuvant chemotherapy (or chemoradiotherapy) completed 6 moths or more before study enrollment is allowed
6. Adequate bone marrow function A. WBCs > 4,000/µL, absolute neutrophil count [ANC]>1,500/µL B. Hemoglobin >9.0 g/dL C. Platelets > 100,000/µL
7. Adequate kidney function (creatinine<1.5 mg/dL)
8. Adequate liver function (bilirubin<1.5 mg/dL [< 2.5 mg/dL for obstructive jaundice with adequately decompressed bile duct obstruction], transaminases levels<3 times the upper normal limit, and serum albumin of >2.5 mg/dL)
9. No serious medical or psychological condition that would preclude study treatment
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Other tumor type than adenocarcinoma
2. Evidence of GI bleeding or GI obstruction
3. Presence or history of CNS metastasis
4. Pregnancy or breastfeeding
5. Other serious illness or medical conditions
6. Axial skeletal radiotherapy within 6 months
7. Neuropathy grade 2 or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | 6 months
  progression-free survival wad defined as the time from the date of enrollment to the date of the first occurrence of objective disease progression or death from any cause, which occur first.

SECONDARY OUTCOMES:
Response rate | 6 months
  Response to chemotherapy will be assessed using RECIST 1.0 criteria.
Toxicities | Up to 24 months
  Toxicities associated chemotherapy will be assessed and categorized using NCI CTCAE v3.0. The types of toxicities and the proportions of patients who experience each toxicity will be described.
overall survival | up to 36 months
  Overall survival is calculated from the date of enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: MJ Kang, MD, MSc, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kang MJ, Lee JL, Kim TW, Lee SS, Ahn S, Park DH, Lee SS, Seo DW, Lee SK, Kim MH. Randomized phase II trial of S-1 and cisplatin versus gemcitabine and cisplatin in patients with advanced biliary tract adenocarcinoma. Acta Oncol. 2012 Sep;51(7):860-6. doi: 10.3109/0284186X.2012.682628. Epub 2012 May 6. PMID 22559158